CLINICAL TRIAL: NCT03353571
Title: A Prospective Evaluation of the Catheter Science C3 "Umbrella Catheter" for Patients With Urinary Retention Due to Bladder Dysfunction (C3 Catheter Study)
Brief Title: A Prospective Evaluation of the Catheter Science C3 "Umbrella Catheter."
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Gaines W. Hammond Jr. MD FACS (Individual)
Responsible Party: Sponsor-Investigator, Dr. Gaines W. Hammond Jr. MD FACS, SPONSOR- INVESTIGATOR, Hammond, Gaines W., Jr., M.D. FACS
Organization: Hammond, Gaines W., Jr., M.D. FACS (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Study # 17/30/08
Record Dates: First submitted 2017-10-24; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Urinary Retention; Urinary Bladder, Neurogenic; Intermittent Catheterization
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Safety and efficacy of the Catheter Science C3 "Umbrella Catheter" in establishing urinary drainage and allowing the control of micturition when indwelling for up to 7 days.
  The reduction in Catheter Acquired Urinary Tract Infection (CAUTI)
  A single arm study design was chosen because there is no alternative treatment to serve as an appropriate control. The C3 catheterizes the bladder with engagement into the bladder neck under the control of the patient or care giver. A Foley catheter, a pre- amendment device, was considered for a control treatment. However, although a Foley catheter is used to establish urinary drainage with close to 100% efficacy, it does not restore voiding function like the C3, and severely impairs activities of daily life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- C3 PATIENT PARTICIPANTS (Other): This single arm prospective study is designed to produce valid scientific evidence regarding safety and efficacy of the C3 in establishing urinary drainage and allowing the control of micturition when indwelling for up to 7 days in patients. The total study population will initially include 50 subjects with open enrollment of additional subjects.
  Interventions: Device: C3 "UMBRELLA CATHETER"

INTERVENTIONS:
Device: C3 "UMBRELLA CATHETER" — The C3 is an alternative method to facilitate bladder drainage in the study population which are using either a foley catheter or Clean Intermittent Catheter technique to drain the bladder.

SUMMARY:
The Catheter Science C3 "Umbrella Catheter" has been developed for management of urinary retention in patients who are either using a Foley or Self Intermittent Catheter. This device is inserted into the bladder in an extended state and once the stylet is removed the device folds into collapsed state. A thread is attached to the device and traverses thru the urethra and is attached to a bobber. With gentle traction on the thread the device engages the bladder neck and the central tube extends which allows for the flow of urine. Once voiding is complete, the thread is released and the device collapses back to the folded state into the bladder. Each voiding cycle is accomplished in a similar fashion. This is a novel technique in which the bladder is catheterized with the device from within the bladder into the bladder neck and urethra. The standard self catheter technique is for placement of a catheter from the outside into the urethra and into the bladder.

DETAILED DESCRIPTION:
Interventional (clinical trial): Participants are assigned prospectively to an intervention or interventions according to a protocol to evaluate the effect of the intervention(s) on biomedical or other health related outcomes.

This single arm, prospective study is designed to produce valid scientific evidence regarding:

1. Safety and efficacy of the Catheter Science C3 "Umbrella Catheter" in establishing urinary drainage and allowing the control of micturition when indwelling for up to 7 days.
2. The reduction in Catheter Acquired Urinary Tract Infection (CAUTI)

A single arm study design was chosen because there is no alternative treatment to serve as an appropriate control. The C3 catheterizes the bladder with engagement into the bladder neck under the control of the patient or care giver. A Foley catheter, a pre- amendment device, was considered for a control treatment. However, although a Foley catheter is used to establish urinary drainage with close to 100% efficacy, it does not restore voiding function like the C3, and severely impairs activities of daily life.

The intrinsic design flaws of a Foley catheter traversing thru the urinary passage which violates the anatomical protective points which help to avoid bacterial contamination. The distal 1/3 portion of the urethra in females is commonly colonized with bacteria. Standard Catheter technique traverses from the outside into the entire length of the urethra to drain the bladder. The standard self catheter flow characteristics are impacted due to the placements of the "eyes" to the catheter lumen. The C3 lumen is open in line with the flow.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Bladder Dysfunction requiring mechanical drainage.
2. Patients with actual urinary retention

Exclusion Criteria:

1. Inability to undergo bladder catheterization (e.g., urethral stricture or history of urethral stricture)
2. Gross hematuria

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Catheterization of the bladder from an antegrade direction with the C3 device. | Measurement of data points are collected sequentially every 7 days up to 28 days.
  The percentage for patients enrolled in the student with the C3 inserted who are able to engage the tubular portion of the device into the bladder neck and urethra from the default position in the bladder with resultant drainage of the bladdder.
The retreat of the C3 back into the bladder from the engaged position | Measurement of data points are collected sequentially every 7 days up to 28 days.
  The percentage of enrolled patients who upon completion of bladder drainage with the engaged tubular portion of the C3 in bladder neck and urethral location retreats back into the default position in the bladder.

SECONDARY OUTCOMES:
Reduction in Catheter Acquired Urinary Tract Infection Rate | Measurement of data points are collected sequentially every 7 days up to 28 days.
  The reduction in Catheter Acquired Urinary Tract Infection (CAUTI) with the C3 "Umbrella Catheter" as compared to the expected incidence with either a Foley Catheter or Self Intermittent Catheter for bladder drainage.

CONTACTS AND LOCATIONS:
Locations (1):
- Watson Clinic Llp, Lakeland, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
LISTED IN STUDY INFORMED CONSENT WITH NAME RECOGNITION WITHHELD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study which is anticipated to be March 2018 for a period of 2 years post completion.
Access Criteria: Access with proper credentials with the patient identifying markers withheld.